CLINICAL TRIAL: NCT01691885
Title: A Randomised, Double-Blind, Placebo-Controlled, Cross-Over, Single-Centre Study to Investigate the Acute Lung Deflation Effects of Fluticasone Furoate/Vilanterol Inhalation Powder 100/25mcg Once Daily on Cardiac Biventricular Function and Arterial Stiffness in Adults With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: RELOVAIR® Lung Deflation Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 116601
Record Dates: First submitted 2012-08-30; First posted 2012-09-25 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A/B (Experimental): Placebo followed by Fluticasone Furoate Vilanterol Combination
  Interventions: Drug: Fluticasone Furoate; Drug: Vilanterol
- B/A (Placebo Comparator): Fluticasone Furoate Vilanterol Combination followed by Placebo
  Interventions: Drug: Fluticasone Furoate; Drug: Vilanterol

INTERVENTIONS:
Drug: Fluticasone Furoate — 100mcg Once daily
  Other Names: RELOVAIR®
Drug: Vilanterol — 25mcg Once daily
  Other Names: RELOVAIR®

SUMMARY:
The primary objective of the study is to test the hypothesis that lung hyperinflation contributes to cardiac dysfunction in COPD and that the treatment of lung deflation with FF/VI Inhalation Powder 100/25 mcg administered once daily (QD) will result in the reversal of this cardiac dysfunction compared with placebo. This will be assessed by measures of right and left global and regional systolic and diastolic cardiac function as assessed using a 30 minute CMR.

A secondary objective will be to investigate the effect of FF/VI inhalation powder 100/25mcg QD on measures of arterial stiffness in the form of pulse wave analysis and distensability in the pulmonary and systemic circulation.

DETAILED DESCRIPTION:
This will be a Phase IIIb, randomised, double-blind, placebo-controlled, cross-over, single-centre study to investigate the acute effects of FF/VI inhalation powder 100/25mcg QD in lung deflation on cardiac biventricular function and arterial stiffness in adults with COPD.

Subjects will visit the clinic a minimum of 4 times over a 28-day period with a further contact which can be either a telephone contact or clinic visit (Visit/Contact 4). A 7-day run-in period will be followed by two 7-day (maximum 14-day) treatment periods separated by a 7(±2) day wash-out period. The first dose of treatment will be taken the day after randomisation. A safety Follow-up contact (either visit or telephone) will occur 7(±2) days post the last treatment day.

Subjects will be prescribed appropriate COPD therapy at the end of Treatment Visit 5, if required. There are no plans to provide the study drug for compassionate use following study completion.

It is planned to have 44 completed evaluable subjects. Subjects who withdraw early will be replaced. In order to ensure 44 evaluable subjects, assuming a 10% protocol deviation rate, 49 subjects will be randomised. The total duration of subject participation, including the follow-up period, will be approximately 36 days.

ELIGIBILITY:
Inclusion Criteria:

* Type of subject: Outpatient.
* Informed consent: Subjects must give their signed and dated written informed consent to participate.
* Gender: Males or females. Female subjects must be post-menopausal or using a highly effective method for avoidance of pregnancy. The decision to include or exclude women of childbearing potential may be made at the discretion of the investigator in accordance with local practice in relation to adequate contraception.
* Age 40 and above
* Smoking history of at least 15 pack years. Previous smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1.
* Established diagnosis of COPD according to ATS/ERS criteria: Subjects with a measured post-albuterol/salbutamol FEV1 less than 70% of predicted normal values; FEV1/FVC ratio after bronchodilator less than 0.7; Post-bronchodilator spirometry will be performed approximately 15 minutes after the subject has self-administered 4 inhalations (i.e., total 400mcg) of salbutamol via an MDI with a valved-holding chamber. The FEV1/FVC ratio and FEV1 percent predicted values will be calculated; MRC SCORE greater than 1
* Residual Volume (RVol) greater than and equal to 20% above predicted value demonstrating evidence of reversibility post bronchodilator of greater than and equal to 7.5% predicted.

Exclusion Criteria:

* Pregnancy: Women who are pregnant or lactating.
* Asthma: Subjects with a current diagnosis of asthma. (Subjects with a prior history of asthma are eligible if they also have a current diagnosis of COPD).
* α1-antitrypsin deficiency: Subjects with known α-1 antitrypsin deficiency as the underlying cause of COPD
* Other respiratory disorders: Subjects with active tuberculosis or lung cancer as well as clinically significant bronchiectasis, sarcoidosis, pulmonary fibrosis, interstitial lung diseases or other active pulmonary diseases. Pulmonary hypertension from causes other than COPD.
* Lung resection or transplantation: Subjects with lung volume reduction surgery within the 12 months prior to Screening or having had a lung transplant or pneumonectomy.
* A moderate/severe COPD exacerbation that has not resolved at least 14 days prior to screening and at least 30 days following the last dose of oral corticosteroids (if applicable).
* Lower respiratory tract infection: Subjects with lower respiratory tract infection that required the use of antibiotics within 6 weeks prior to screening.
* Pulmonary Rehabilitation: Patients to be excluded if they have been in the acute phase of pulmonary rehabilitation in the 4 weeks prior to screening
* Current severe heart failure (New York Heart Association class IV) [New York HeartAssociation, 1994]. Subjects will also be excluded if they have a known ejection fraction of less than 30%.
* Abnormal and clinically significant 12-lead ECG
* Other systemic inflammatory conditions associated with chronic inflammation in the opinion of the investigator (e.g. rheumatoid arthritis, connective tissue disorders and Inflammatory Bowel Disease)
* Other significant diseases / abnormalities: Any life-threatening condition with life expectancy greater than 1 year, other than vascular disease or COPD, that might prevent the subject from completing the study.
* Coronary Artery Bypass Grafting (CABG) in the 6 months prior to screening.
* Myocardial infarction, cerebrovascular event or coronary artery intervention other than CABG in the 1 month prior to screening.

Inclusion of these patients with events over 1 month prior to screening will be based on physician's judgment.

* History of malignancy within the past 5 years, other than non-melanoma skin cancer.
* End stage chronic renal disease: Subjects will be excluded if on renal replacement therapy (hemodialysis or peritoneal). Drug/food allergy: Subjects with a history of hypersensitivity to any of the study medications (e.g. beta-agonists, corticosteroid) or components of the inhalation powder (e.g. lactose, magnesium stearate). In addition, patients with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates the subject's participation will also be excluded.
* Drug/alcohol abuse: Subjects with a known or suspected history of alcohol or drug abuse within the last 2 years.
* Oxygen therapy: Subjects receiving treatment with long-term oxygen therapy (LTOT) or nocturnal oxygen therapy required for greater than 12 hours a day. Oxygen should not be initiated during the trial.
* Questionable validity of consent: Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study or the potential compliance to study procedures.
* Additional medication: Use of an investigational device or investigational drug within 30 days or 5 half-lives (whichever is longer) preceding the first dose of study medication.
* Use of the following medications is not permitted within the following timeframes: Prohibited Treatment: Depot corticosteroids, Time: 12 weeks; Prohibited Treatment: Cytochrome P450 3A4 strong inhibitors including but not limited to antiretrovirals (protease inhibitors) (e.g., indinavir, nelfinavir, ritonavir, saquinavir, atazanavir); imidazole and triazole anti- fungals (e.g., ketaconazole, itraconazole, voriconazole); clarithromycin, telithromycin, troleandomycin, mibefradil, cyclosporin, nefazodone, Time: 6 weeks, Grapefruit is allowed up to Visit 1, then limited to no more than one glass of grapefruit juice (250 mL/8 ounces) or one grapefruit per day (The use of cytochrome p450 3A4 inhibitors and inducers in the presence of significant liver impairment will result in the participant being excluded from the trial); Prohibited Treatment: Systemic, oral, parenteral (intra-articular) corticosteroids, Time: 30 days; Prohibited Treatment: Antibiotics, Time: 6 weeks; Prohibited Treatment: Inhaled corticosteroids, Time: 2 weeks; Inhaled ICS/LABA combination products, Time: 2 weeks; Prohibited Treatment: Long-acting anticholinergics (e.g., tiotropium), Time: 4 days; Prohibited Treatment: PDE-4 inhibitors (e.g., roflumilast), Time: 1 week; Prohibited Treatment: Oral leukotriene inhibitors (e.g., zafirlukast, montelukast, zileuton), Time: 48 hours; Prohibited Treatment: Inhaled long acting beta2-agonists (LABA) (e.g., salmeterol), Time: 48 hours; Prohibited Treatment: Oral beta-agonists, Time: 48 hours; Prohibited Treatment: Inhaled sodium cromoglycate or nedocromil sodium, Time: 24 hours; Prohibited Treatment Ipratropium/albuterol (salbutamol) combination product, Time: 6 hours; Prohibited Treatment: Short-acting anti-cholinergics (e.g., ipratropium bromide), Time: 6 hours (ipratropium will be supplied for rescue during the study, in inhaled or nebulized form); Prohibited Treatment: Theophylline preparations, Time: 48 hours; Prohibited Treatment: Inhaled short-acting beta2-agonists, Time: 6 hours (albuterol/salbutamol will be supplied for rescue during the study, in inhaled or nebulized form)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Khanji MY, Stone IS, Boubertakh R, Cooper JA, Barnes NC, Petersen SE. Chronic Obstructive Pulmonary Disease as a Predictor of Cardiovascular Risk: A Case-Control Study. COPD. 2020 Feb;17(1):81-89. doi: 10.1080/15412555.2019.1694501. Epub 2019 Dec 13. PMID 31833441
- [Derived] Stone IS, Barnes NC, James WY, Midwinter D, Boubertakh R, Follows R, John L, Petersen SE. Lung Deflation and Cardiovascular Structure and Function in Chronic Obstructive Pulmonary Disease. A Randomized Controlled Trial. Am J Respir Crit Care Med. 2016 Apr 1;193(7):717-26. doi: 10.1164/rccm.201508-1647OC. PMID 26550687
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 116601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116601 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: At Visit 1a, participants who met the eligibility criteria stopped their respiratory medication in preparation for their lung volume assessment at screening Visit 1b. At Visit 1b, participants entered a 7(plus or minus 3) day Run-in Period. Overall study duration, following Screening to Follow-up, was 36 days up to a maximum of 54 days.
Groups:
- Placebo Then FF/VI: Participants entering Treatment Period 1 received matching placebo once daily (QD), each morning via a dry powder inhaler (DPI) for a period of 7 days, up to a maximum of 14 days. Following Treatment Period 1, participants entered a washout period for 7 days, up to a maximum of 9 days. Following the washout period participants entered Treatment Period 2 and received Fluticasone Furoate/Vilanerol (FF/VI) 100/25 micrograms (µg), QD, each morning via a DPI for 7 days, up to a maximum of 14 days.
- FF/VI Then Placebo: Participants entering Treatment Period 1 received FF/VI 100/25 µg QD, each morning via a DPI for a period of 7 days, up to a maximum of 14 days. Following Treatment Period 1, participants entered a washout period for 7 days, up to a maximum of 9 days. Following the washout period, participants entered Treatment Period 2 and received matching placebo QD, each morning via a DPI for 7 days, up to a maximum of 14 days.
Period: Treatment Period 1(7-14 Days)
Arm/Group | Placebo Then FF/VI | FF/VI Then Placebo
Started | 22 | 23
Completed | 21 | 22
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Washout Period (7-9 Days)
Arm/Group | Placebo Then FF/VI | FF/VI Then Placebo
Started | 21 | 22
Completed | 21 | 21
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Treatment Period 2 (7-14 Days)
Arm/Group | Placebo Then FF/VI | FF/VI Then Placebo
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Per Protocol Population: All participants received placebo or FF/VI 100/25 µg in either of the two treatment periods QD, each morning from a DPI. Treatment periods lasted 7 days up to a maximum of 14 days for each period. The two treatments were separated by a wash out period of 7 days, up to a maximum of 9 days.
Arm/Group | Per Protocol Population
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 28
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 6
  White - White/Caucasian/European Heritage | 39

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Right Ventricular End Diastolic Volume Index (RVEDVI) at the End of the Overall Treatment Period
Description: RVEDVI is a measure of the volume of blood in the right ventricle at the end of diastole, normalized over body surface area and was measured using Cardiac Magnetic Resonance (CMR) imaging. RVEDVI is calculated as the right ventricular end diastolic volume (RDEDV) divided by the body surface area (BSA). The change from Baseline in RVEDVI was analyzed using a mixed model analysis with period, treatment group, and Baseline RVEDVI fitted as fixed effects and participants fitted as a random effect. The Baseline is defined as the assessment performed pre-dose at Day 1 of Treatment Period 1. The change from Baseline is calculated as the RVEDVI value at the end of each treatment period minus the Baseline value. The Per Protocol (PP) Population was comprised of all participants in the modified intent-to-treat (mITT) Population not identified as having deviations considered to impact the primary efficacy analysis.
Time Frame: Baseline and end of Treatment Period (7 days)
Population: PP Population. Only those participants available at the specified time points were analyzed
Measure: Least Squares Mean (Standard Error); unit: Milliliter per meter square (mL/m^2)
Groups:
- Placebo: Participants received matching placebo once daily (QD), each morning via a dry powder inhaler (DPI) for a period of 7 days, up to a maximum of 14 days during one of the two Treatment Periods. Participants that received placebo in Treatment Period 1, crossed over after the washout period to receive FF/VI 100/25 μg during Treatment Period 2. Participants that received FF/VI 100/25 μg during Treatment Period 1, crossed over after the washout period to receive placebo during Treatment Period 2.
- FF/VI: Participants received FF/VI 100/25 μg QD, each morning via a DPI for a period of 7 days, up to a maximum of 14 days during one of the two Treatment Periods. Participants that received FF/VI 100/25 μg in Treatment Period 1, crossed over after the washout period to receive placebo during Treatment Period 2. Participants that received placebo during Treatment Period 1, crossed over after the washout period to receive FF/VI 100/25 μg during Treatment Period 2.
Arm/Group | Placebo | FF/VI
Number analyzed (Participants) | 41 | 43
Milliliter per meter square (mL/m^2) | -0.47 (1.393) | 5.35 (1.365)
Statistical Analysis 1: Comparison: Placebo vs FF/VI; Test type: Superiority or Other; p < 0.001, ANCOVA; Analysis was performed using an ANCOVA model with covariates of treatment, baseline, period and subject as a random effect; Mean Difference (Final Values) = 5.83, 95% CI 2-sided [2.74 to 8.91]

ADVERSE EVENTS:
Time Frame: On treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment and up to the end of treatment (Study Day 23)
Arm/Group | Placebo | FF/VI
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/44
Other Adverse Events (participants affected / at risk) | 2/43 | 2/44
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=43) | FF/VI (N=44)
Headache (Nervous system disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.